CLINICAL TRIAL: NCT05743530
Title: Effect of Perioperative Neurostimulation in Patients Undergoing Whipple Operation (Pancreaticoduodenectomy) on Acute Postsurgical Inflammatory Response [ENSWAPI-trial]
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENSWAPI
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Pancreaticoduodenectomy
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS - transcutaneous electrical nerve stimulation (Experimental)
  Interventions: Device: TENS - transcutaneous electrical nerve stimulation
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Device: TENS - transcutaneous electrical nerve stimulation — Pre-operative day 1 till postoperative day 14.
  Arms: TENS - transcutaneous electrical nerve stimulation
Other: Placebo — Pre-operative day 1 till postoperative day 14.
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to test whether electrical stimulation of the vagus nerve via a device placed on the top of the external ear can reduce the postoperative inflammatory reaction after Whipple's surgery (pancreatoduodenectomy).

DETAILED DESCRIPTION:
Following surgery, inflammation normally is a balanced event, which is resolved in a timely manner. But, disrupted immune regulation can result in continuous proinflammatory cytokine activity and excessive or chronic inflammation. In the case of major surgical interventions, the inflammatory reaction is not limited to the area of surgery, but takes place systemically via various mediators. The cytokines IL-1, TNF-α and IL-6, which are formed by the leukocytes, are responsible for associated clinical symptoms like fever, fatigue and general feeling of illness. By crossing the blood-brain barrier, IL-6 initiates the synthesis of prostaglandin E2 (PGE2), and IL-6 also facilitates energy mobilizations in muscle and fat tissue. The release of acute phase proteins from the hepatocytes of the liver is also effected via cytokines. These include fibrinogen and C-reactive protein (CRP), which are involved in the removal of entered microorganisms with opsonization and complement fixation. However, if too many of these cytokines are present or if they are released for prolonged periods, this can lead to an intensified inflammatory process, which is also called systemic inflammatory response syndrome (SIRS) if certain criteria are met. These criteria include systemic activation of the coagulation cascade, disseminated intravascular coagulation (DIC), Acute Respiratory Distress Syndrome (ARDS) and Multi Organ Failure (MOF). In the worst case, this ends with the patient's death. In order to avoid destruction by one's own immune system, pro-inflammatory mediators are only released for a short time. In addition, the organism forms anti-inflammatory mediators such as Transforming Growth Factor Beta (TGF-ß) and IL-10, which is formed by the TH2 subtype of CD4 positive T lymphocytes. They counteract the inflammatory process by downregulating the immune response and thus limiting the destruction of the tissue.

A well-functioning immune system is essential for surgery. The interaction of inflammation and anti-inflammation ensures the destruction of the destroyed tissue and prevents penetrating microorganisms from developing an infection. An excessive pro-inflammatory reaction can lead to a SIRS, a possibly reactive strong post-operative immunosuppression facilitates the penetration of pathological microorganisms and thus predisposes to infection. Unfortunately, postoperative infectious and non-infectious postoperative complications do occur in spite of preventive treatment with antibiotics immediately before or during surgical treatment and have so far been treated upon their occurrence during the postoperative recovery period.

An analysis on postoperative morbidity associated with inflammation in pancreatic surgery (own database (n=275)) showed the development of postoperative sepsis in 4% (n=11), which had an abdominal focus in 2.9% (n=8) and other localizations in 1.1% (n=3). Postoperative pneumonia has been reported to occur after pancreatic resection in 1-6% of cases and has been associated with both pancreatic fistula and delayed gastric emptying (DGE), and has been reported to be associated with a very high 90-day-mortality [6]. IL-6 is a major mediator of inflammation, and it is important to elucidate that IL-6 is part of a complex, interdepending network of cytokines released in inflammatory conditions [7]. In healthy adults, IL-6 concentrations in the plasma are <10 pg/ml [8]. IL-6 is particularly important in chronic inflammatory conditions such as rheumatoid arthritis, inflammatory bowel disease, Castlemann's disease, haematopoietic diseases and after physical stress such as surgery or chemotherapy. Increased levels of serum and/or tumor IL-6 are also seen in a number of malignant conditions, both haematopoietic malignancies and solid tumors including breast, cervical, esophageal, head-and-neck, ovarian, prostate, colorectal, pancreatic, hepatocellular, gall bladder, non-small-cell lung cancer and multiple myeloma, reflecting the immunological involvement in cancer. Several studies have shown IL-6 to be a prognostic indicator of survival as well as predictive in response to therapy in many types of cancer [9, 10]. A high IL-6 level is generally associated with a poorer outcome and with more severe symptoms in regards to cancer as well as the development of anti-cancer drug resistance [11, 12].

Endogenous mechanisms that prevent or neutralize excessive proinflammatory reactions could lead to novel therapeutic options.

Transcutaneous electrical neurostimulation (TENS) is a non-invasive physiotherapeutic resource for pain management, but evidence on the effectiveness of this device at reducing proinflammatory cytokines in the blood is unclear.

TENS is a strategy that allows for interaction with the peripheral vascular system or with the autonomic nervous system.

The vagus nerve is the main nerve of the parasympathetic division of the autonomic nervous system. The vagus nerve regulates metabolic homeostasis by controlling heart rate, gastrointestinal motility and secretion, pancreatic endocrine and exocrine secretion, hepatic glucose production, and many other visceral functions over the brainstem. In addition, afferent and efferent branches of the vagus nerve are part of a neural reflex mechanism (the inflammatory reflex) that controls innate immune responses and inflammation during pathogen invasion and tissue injury [1, 2, 3]. Innate immune responses are activated by pathogen-associated and danger-associated molecular patterns. Activation of downstream signaling cascades results in increased production and release of tumor necrosis factor (TNF), IL-6 and other proinflammatory cytokines. These are implicated in extracellular pathogen clearance, vasodilatation, neutrophil recruitment, increased vascular permeability and induction of acute-phase proteins, such as C-reactive protein (CRP), and coagulation molecules. Proinflammatory progression is balanced by the release of IL-10, TGF-ß and other anti-inflammatory molecules.

Communication between the immune system and the brain is vital for controlling inflammation by the inflammatory reflex (the afferent vagus nerve signalling, which is activated by cytokines or pathogen-derived products, is functionally associated with efferent vagus nerve-mediated regulation of proinflammatory cytokine production and inflammation) [2, 3]. The inflammatory reflex is a physiological mechanism through which the nervous system maintains immunologic homeostasis by modulating innate and adaptive immunity. The absence of this inflammatory reflex leads to excessive immune responses and cytokine toxicity. It could be shown that the severity of collagen-induced arthritis can be reduced by neurostimulation of the cholinergic anti-inflammatory pathway, supporting the rationale for testing this approach in human inflammatory disorders [4]. Koopman et al. have shown that the vagus nerve stimulation (up to four times daily) for the reduction of the frequency of epileptic seizures had an effect also on the activity of rheumatoid arthritis. The vagus nerve stimulation significantly inhibited the TNF production for up to 84 days [5]. These results establish that vagus nerve stimulation modulates TNF production and reduces inflammation in humans. Gürgen et al. found that distinctive decreases of pro-inflammatory cytokines observed in the dermis in the vagus nerve stimulation group suggest that TENS shortened the healing process by inhibiting the inflammation phase in an animal model on wound healing in terms of the expression levels of pro-inflammatory cytokines [13]. We intend to investigate the effect of perioperative vagus nerve stimulation by application of the Neurostimulator V by Ducest in patients undergoing Whipple operation (pancreaticoduodenectomy).

ELIGIBILITY:
Inclusion Criteria:

* Patients (male/female) scheduled for Whipple procedure (pancreaticoduodenectomy)
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent must be available before enrolment in the trial

Exclusion Criteria:

* Patients < 18 and > 90 years of age
* Simultaneous participation in other clinical trials
* Pregnancy
* Current infection
* Hemophilia
* Psoriasis vulgaris
* Pacemaker, implanted cardioverter defibrillator, cardiac resynchronization therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
IL-6 levels change | Baseline and postoperative day 1
  IL-6 levels change between baseline and postoperative day 1. Baseline is defines as the serum concentration IL-6 at 24h prior to surgery

SECONDARY OUTCOMES:
Post surgical inflammatory response (IL-1) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (IL-6) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (IL-8) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (IL-13) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (IL-10) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (IL-18) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (TLF-alpha) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (IFN-gamma) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (IL-1-beta) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (Serum Zonulin) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (LPS) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (Serum Ketone) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (HBA1c) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (NH3) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
Post surgical inflammatory response (GLP-1) | before surgery, day 1 and day 4 after surgery
  measurement of several cytocine levels over time
AST | Before surgery; daily between day 1 and day 7, on day 14 and day 90 after surgery
  routine clinical parameters
AP | Before surgery; daily between day 1 and day 7, on day 14 and day 90 after surgery
  routine clinical parameters
GGT | Before surgery; daily between day 1 and day 7, on day 14 and day 90 after surgery
  routine clinical parameters
ALT | Before surgery; daily between day 1 and day 7, on day 14 and day 90 after surgery
  routine clinical parameters
LDH | Before surgery; daily between day 1 and day 7, on day 14 and day 90 after surgery
  routine clinical parameters
CK | Before surgery; daily between day 1 and day 7, on day 14 and day 90 after surgery
  routine clinical parameters
Bilirubin | Before surgery; daily between day 1 and day 7, on day 14 and day 90 after surgery
  routine clinical parameters
CRP | Before surgery; daily between day 1 and day 7, on day 14 and day 90 after surgery
  routine clinical parameters
Procalcitronin | Before surgery; daily between day 1 and day 7, on day 14 and day 90 after surgery
  routine clinical parameters
VOCs | 1x preoperative and on postoperative day 4
Microbiome analysis | 1x preoperative and on postoperative day 4
  S-16 based microbiomanalysis (oral swap)
Microbiome analysis | 1x interoperatively
  Pancreatic fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Allgemein,- Viszeral,- Transplantationschirurgie LKH Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tracey KJ. The inflammatory reflex. Nature. 2002 Dec 19-26;420(6917):853-9. doi: 10.1038/nature01321. PMID 12490958
- [Background] Tracey KJ. Reflex control of immunity. Nat Rev Immunol. 2009 Jun;9(6):418-28. doi: 10.1038/nri2566. PMID 19461672
- [Background] Pavlov VA, Tracey KJ. The vagus nerve and the inflammatory reflex--linking immunity and metabolism. Nat Rev Endocrinol. 2012 Dec;8(12):743-54. doi: 10.1038/nrendo.2012.189. PMID 23169440
- [Background] Levine YA, Koopman FA, Faltys M, Caravaca A, Bendele A, Zitnik R, Vervoordeldonk MJ, Tak PP. Neurostimulation of the cholinergic anti-inflammatory pathway ameliorates disease in rat collagen-induced arthritis. PLoS One. 2014 Aug 11;9(8):e104530. doi: 10.1371/journal.pone.0104530. eCollection 2014. PMID 25110981
- [Background] Koopman FA, Chavan SS, Miljko S, Grazio S, Sokolovic S, Schuurman PR, Mehta AD, Levine YA, Faltys M, Zitnik R, Tracey KJ, Tak PP. Vagus nerve stimulation inhibits cytokine production and attenuates disease severity in rheumatoid arthritis. Proc Natl Acad Sci U S A. 2016 Jul 19;113(29):8284-9. doi: 10.1073/pnas.1605635113. Epub 2016 Jul 5. PMID 27382171
- [Background] Nagle RT, Leiby BE, Lavu H, Rosato EL, Yeo CJ, Winter JM. Pneumonia is associated with a high risk of mortality after pancreaticoduodenectomy. Surgery. 2017 Apr;161(4):959-967. doi: 10.1016/j.surg.2016.09.028. Epub 2016 Nov 8. PMID 27836210
- [Background] Patel SA, Gooderham NJ. IL6 Mediates Immune and Colorectal Cancer Cell Cross-talk via miR-21 and miR-29b. Mol Cancer Res. 2015 Nov;13(11):1502-8. doi: 10.1158/1541-7786.MCR-15-0147. Epub 2015 Jul 16. PMID 26184038
- [Background] Song M, Kellum JA. Interleukin-6. Crit Care Med. 2005 Dec;33(12 Suppl):S463-5. doi: 10.1097/01.ccm.0000186784.62662.a1. No abstract available. PMID 16340422
- [Background] Johnson DE, O'Keefe RA, Grandis JR. Targeting the IL-6/JAK/STAT3 signalling axis in cancer. Nat Rev Clin Oncol. 2018 Apr;15(4):234-248. doi: 10.1038/nrclinonc.2018.8. Epub 2018 Feb 6. PMID 29405201
- [Background] Koca YS, Bulbul M, Barut I. The Diagnostic Roles of Cytokines in Hepatobiliary Cancers. Biomed Res Int. 2017;2017:2979307. doi: 10.1155/2017/2979307. Epub 2017 Dec 19. PMID 29410961
- [Background] Vainer N, Dehlendorff C, Johansen JS. Systematic literature review of IL-6 as a biomarker or treatment target in patients with gastric, bile duct, pancreatic and colorectal cancer. Oncotarget. 2018 Jul 3;9(51):29820-29841. doi: 10.18632/oncotarget.25661. eCollection 2018 Jul 3. PMID 30038723
- [Background] Angele MK, Faist E. Clinical review: immunodepression in the surgical patient and increased susceptibility to infection. Crit Care. 2002 Aug;6(4):298-305. doi: 10.1186/cc1514. Epub 2002 May 24. PMID 12225603
- [Background] Gurgen SG, Sayin O, Cetin F, Tuc Yucel A. Transcutaneous electrical nerve stimulation (TENS) accelerates cutaneous wound healing and inhibits pro-inflammatory cytokines. Inflammation. 2014 Jun;37(3):775-84. doi: 10.1007/s10753-013-9796-7. PMID 24357416
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Background] Trefz P, Rosner L, Hein D, Schubert JK, Miekisch W. Evaluation of needle trap micro-extraction and automatic alveolar sampling for point-of-care breath analysis. Anal Bioanal Chem. 2013 Apr;405(10):3105-15. doi: 10.1007/s00216-013-6781-9. Epub 2013 Feb 7. PMID 23388692